CLINICAL TRIAL: NCT00636194
Title: Product Performance of Bausch & Lomb Multi-Purpose Solution Compared to Alcon Opti-Free Replenish Multi-Purpose Solution When Used With Silicone Hydrogel Contact Lenses Worn on a Daily Wear Basis
Brief Title: Comparative Performance of a Bausch & Lomb Multipurpose Solution and Alcon OptiFree Replenish Multipurpose Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 562
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Results first posted 2011-02-15 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Adverse Effect of Contact Lens Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- B&L Multipurpose solution (Experimental): Bausch & Lomb Multipurpose Contact Lens Solution
  Interventions: Device: Bausch & Lomb Multipurpose Solution
- Alcon Multipurpose Solution (Active Comparator): Alcon OptiFree Replenish Multipurpose Contact Lens Solution
  Interventions: Device: Alcon OptiFree Replenish Multipurpose Solution

INTERVENTIONS:
Device: Bausch & Lomb Multipurpose Solution — daily care of contact lenses
  Arms: B&L Multipurpose solution
Device: Alcon OptiFree Replenish Multipurpose Solution — daily care for contact lenses
  Arms: Alcon Multipurpose Solution

SUMMARY:
To evaluate the product performance of a Bausch & Lomb Multipurpose solution when compared to Alcon OptiFree Replenish Multipurpose Solution

ELIGIBILITY:
Inclusion Criteria:

* Subjects are adapted wearers of silicone hydrogel contact lenses
* VA correctable to 0.3 LogMAR or better (driving vision)
* Clear central cornea
* Subject uses a lens care system on a regular basis

Exclusion Criteria:

* Systemic disease affecting ocular health
* Using systemic or topical medications
* wear a monovision, multifocal or toric contact lenses
* Any grade 2 or greater slit lamp findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohinder Merchea, OD, PhD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Laser Focus Sdn Bhd, Vision Correction Centre, Jalan Kuning, Tamn Pelangi, Johor Bahru, Malaysia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 361 subjects (722 eyes) who are currently adapted silicone hydrogel contact lens wearers and are habitually using a lens care product for disinfecting lenses, were enrolled in this 2-Week study at approximately 14 investigative sites in Asia. Study start date was 2/16/2008 and last subject exited on 3/17/2008.
Pre-assignment Details: Fourteen Investigators enrolled 361 subjects in the study. Of these subjects, 347 successfully completed the study, 3 discontinued and 11 were ineligible at baseline, but were dispensed study materials
Period: Overall Study
Arm/Group | B&L Multipurpose Solution | Alcon Multipurpose Solution
Started | 175 | 175
Completed | 172 | 175
Not Completed | 3 | 0
Not completed — Study related symptoms and complaints | 1 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | B&L Multipurpose Solution | Alcon Multipurpose Solution | Total
Number analyzed (Participants) | 175 | 175 | 350
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 175 | 175 | 350
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 121 | 246
  Male | 50 | 54 | 104
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 175 | 175 | 350

OUTCOME MEASURES:

1. Primary Outcome: Subjective Assessment of Comfort and Cleanliness
Description: Scale from 0-100 for each eye where 100=most favorable rating and 0=the least favorable rating.
Time Frame: 7 days
Population: All eyes
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: eyes
Arm/Group | B&L Multipurpose Solution | Alcon Multipurpose Solution
Number analyzed (Participants) | 174 | 175
Number analyzed (eyes) | 348 | 350
Scores on a scale
  Cleanliness upon insertion | 89.71 (14.52) | 89.26 (14.52)
  Comfort upon insertion | 87.45 (15.56) | 86.63 (15.56)
  Cleanliness at end of day | 82.98 (18.54) | 82.34 (18.54)
  Comfort at end of day | 80.14 (19.41) | 79.60 (19.41)

2. Secondary Outcome: Symptoms and Complaints
Description: Scores on a scale from 0 to 100, with 100 being the most favorable. Eyes with multiple unscheduled visits in a visit category were counted once for their lowest score.
Time Frame: 2 weeks
Population: All eligible, dispensed eyes
Measure: Mean (Standard Deviation); unit: Score on a scale
Units Other Than Participants: eyes
Arm/Group | B&L Multipurpose Solution | Alcon Multipurpose Solution
Number analyzed (Participants) | 173 | 175
Number analyzed (eyes) | 346 | 350
Score on a scale
  Comfort | 85.4 (14.7) | 86.1 (13.1)
  End of day comfort | 79.2 (16.7) | 79.3 (15.1)
  Burning/stinging upon insertion | 87.0 (18.7) | 88.9 (14.8)
  Irritation | 86.4 (18.7) | 88.2 (14.6)
  Itching | 89.2 (16.6) | 90.3 (13.2)
  Dryness | 80.6 (16.6) | 81.9 (15.7)
  Redness | 89.2 (15.8) | 90.0 (12.7)
  Vision | 89.8 (13.1) | 89.4 (12.5)
  Lens cleanliness | 86.6 (14.6) | 86.9 (13.1)
  Lens handling | 90.8 (11.4) | 90.4 (11.0)

3. Secondary Outcome: Graded Slit Lamp Findings > Grade 2
Description: Grade none (no findings) - grade 4 (severe findings). Eyes in the Test group were compared with eyes in the Control group. Slit lamp finding greater than Grade 2.
Time Frame: 2 week follow-up visit
Population: All dispensed, completed eyes
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | B&L Multipurpose Solution | Alcon Multipurpose Solution
Number analyzed (Participants) | 172 | 175
Number analyzed (eyes) | 344 | 350
eyes
  Epithelial edema | 0 | 0
  Epithelial microcysts | 0 | 0
  Corneal staining | 3 | 0
  Limbal injection | 0 | 0
  Bulbar injection | 0 | 0
  Superior tarsal conjunctival abnormalities | 0 | 0
  Corneal neovascularization | 0 | 0
  Corneal infiltrates | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | B&L Multipurpose Solution | Alcon Multipurpose Solution
Serious Adverse Events (participants affected / at risk) | 0/175 | 0/175
Other Adverse Events (participants affected / at risk) | 0/175 | 0/175

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.

Prior to publication or presentation, a copy of the final text should be forwarded by the Investigator(s) to the Sponsor or its designee, for comment.